CLINICAL TRIAL: NCT04010994
Title: Treatment of Patients With Optic Nerve Damage Patients Using Electrostimulation: a Home Stimulation Study
Brief Title: Treatment of Patients With Optic Nerve Damage Patients Using Electrostimulation
Acronym: HomeStim
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Head of Institute, Professor, University of Magdeburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StimulationMagd
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Glaucoma; Electrical Stimulation; Home Treatment
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rtACS (Other): repetitive transorbital ACS
  Interventions: Procedure: Transorbital electrical stimulation

INTERVENTIONS:
Procedure: Transorbital electrical stimulation — Transorbital ACS using 8-12 Hz with 0,5-1,5 mA Intensity, during the first two weeks 1/day, after 2/week for 10 weeks, as a home treatment

SUMMARY:
The aim of the present study is to investigate the possibilities of visual field enhancement with electrical stimulation (ES) as a home stimulation method, in a total of 50 patients with optical neuropathy, who have already been treated with ES in the past.

Furthermore, factors responsible for response variability and treatment effectiveness are also explored: (i) the role of mental stress (or stress resilience), (ii) the status of biomarkers, such as the systemic stress hormone levels and blood supply to the eye and brain (specifically vascular dysregulation) and (iii) the influence of personality, anxiety, depression and lifestyle. The study serves to further validate this ES procedure for the treatment of visual impairment. Specifically, better efficacy, better compliance, lowest response variability are expected after long-term home use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma, disease duration at least 6 months
* stable visual field defect across baseline measurement (subjects with spontaneous fluctuations and recovery of vision excluded)
* presence of residual vision and detectable gradual transition between the intact and the absolutely blind part of the visual field according to evaluation of the clinician
* best corrected visual acuity at least 0.4 (20/50 Snellen) or better

Exclusion Criteria:

* autoimmune diseases in the acute stage
* neurological and mental diseases
* diabetic retinopathy
* addictions
* hypertension (maximum 160/100 mmHg)
* retinitis pigmentosa-
* pathological nystagmus
* non-distant tumors or recurrent tumors
* photosensitivity
* pregnancy
* electric or electronic implants (e.g. heart pacemaker)
* metal implants in the eyes or head (with the exception of dental prosthesis or shunts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual field size | 3 months
  Static perimetry and high resolution perimetry will be used to measure the visual field sizes

SECONDARY OUTCOMES:
EEG connectivities in the visual system | 3 months
  EEG recordings will be done using 128 channels, power spectra will be determined
Level of vascular regulation/dysregulation in the eye | 3 months
  Dynamic vessel analysis will be used the measure blood flow in the eye

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Psychology, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available without restriction
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication
Access Criteria: Contact to the Principal investigator

REFERENCES:
- [Background] Gall C, Schmidt S, Schittkowski MP, Antal A, Ambrus GG, Paulus W, Dannhauer M, Michalik R, Mante A, Bola M, Lux A, Kropf S, Brandt SA, Sabel BA. Alternating Current Stimulation for Vision Restoration after Optic Nerve Damage: A Randomized Clinical Trial. PLoS One. 2016 Jun 29;11(6):e0156134. doi: 10.1371/journal.pone.0156134. eCollection 2016. PMID 27355577